CLINICAL TRIAL: NCT06289751
Title: Neoadjuvant Chemotherapy Plus Cadunilizumab Followed by Extrafascial Hysterectomy for FIGO Stage IB2 Cervical Cancer: a Multicenter, Single-arm, Phase 2 Trial.
Brief Title: Neoadjuvant Chemoimmunotherapy and Extrafascial Hysterectomy for IB2 Cervical Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tongji Hospital (Other)
Collaborators: The First Affiliated Hospital of China University of Science and Technology (Anhui Provincial) (Other); Women's Hospital School Of Medicine Zhejiang University (Other); Southwest Hospital, China (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Sichuan Cancer Hospital and Research Institute (Other); Qilu Hospital of Shandong University (Other); Beijing Friendship Hospital (Other); Tianjin Medical University (Other); West China Second University Hospital (Other); Xiangya Hospital of Central South University (Other); Gansu Provincial Maternal and Child Health Care Hospital (Other); Zhejiang Cancer Hospital (Other); Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Gang Chen (101199), Professor, Tongji Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NACI-CerV-004
Record Dates: First submitted 2024-02-22; First posted 2024-03-04 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Cervical Cancer; Neoadjuvant Chemoimmunotherapy; Radical Hysterectomy; Extrafascial Hysterectomy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Conization

STUDY DESIGN:
Intervention Model Description: a multicentre, single-arm, phase 2 trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant chemoimmunotherapy for ⅠB2 cervical cancer (Experimental): neoadjuvant chemotherapy + Cadonilimab + Radical hysterectomy/Extrafascial hysterectomy
  Interventions: Drug: Cadonilimab; Drug: Paclitaxel-albumin; Drug: Cisplatin; Procedure: Extrafascial hysterectomy; Procedure: Radical hysterectomy; Procedure: Cone biopsy

INTERVENTIONS:
Drug: Cadonilimab — 10 mg/kg (body weight), 60 min, IV. Repeat every 3 weeks for a total of 3 cycles
  Other Names: Cadonilimab Injection; AK104
Drug: Paclitaxel-albumin — 260 mg/m2 for 30 min. Repeat every 3 weeks for a total of 3 cycles.
  Other Names: Injectable paclitaxel (albumin bound)
Drug: Cisplatin — 75-80 mg/m2, IV, 1 mg/min. Repeat every 3 weeks for a total of 3 cycles.
  Other Names: Cisplatin injection
Procedure: Extrafascial hysterectomy — Extrafascial hysterectomy + pelvic lymphadenectomy (or SLN mapping) (For participants who meet ConCerv criteria)
Procedure: Radical hysterectomy — Radical hysterectomy + pelvic lymphadenectomy ± para-aortic lymphadenectomy (or SLN mapping) (For participants who do not meet ConCerv criteria)
Procedure: Cone biopsy — Cold knife conization (CKC) (For participants with tumor size ≤2 cm after 3 cycles of chemo-immunotherapy)

SUMMARY:
This study is an exploratory clinical trial to investigate the feasibility of neoadjuvant chemoimmunotherapy plus extrafascial hysterectomy and pelvic lymph node dissection in patients with stage IB2 (2018 FIGO) cervical cancer and to observe the response rate to treatment, adverse effects and complications, and to assess the survival rate of patients.

DETAILED DESCRIPTION:
In China, cervical cancer is the malignant tumor of the female reproductive tract with the highest incidence rate, and there will be about 112,000 new cases of cervical cancer and 14,000 deaths in China in 2022, with the number of incidence cases accounting for 1/5 of the global total. In recent years, with the early detection of cervical cancer and the wide application of HPV vaccine, more and more patients have been diagnosed at an early stage, which has prompted researchers to conduct in-depth studies and investigations into the treatment of early cervical cancer. to conduct in-depth studies and investigations. For a long time, the standard treatment for early-stage cervical cancer has been wide radical hysterectomy combined with pelvic lymph node dissection, with satisfactory results and 5-year overall survival rates ranging from 73% to 98%. The core of radical hysterectomy is wide hysterectomy, which ensures complete removal of the cervix and uterine body and achieves negative margins. However, this procedure is associated with high complications. In addition to ligamentous penetration, there are important neurovascular vessels in the parietal tissues, which will increase the risk of intraoperative complications such as bleeding, nerve injury, urinary tract and bowel injury, etc. Postoperative complications such as urinary retention, urinary incontinence, defecation difficulties, constipation, and sexual dysfunction may also occur in the immediate and long-term future, which will cause serious problems to the patient's quality of life, especially to the family harmony and social role of young patients. Realization brings serious disturbances.

It has been controversial whether radical hysterectomy is necessary to remove paracervical tissue in early-stage cervical cancer. Studies have reported that the probability of paracervical infiltration is less than 1% in patients with tumors less than 2 cm in diameter, no lymphovascular invasion, and no metastasis in the pelvic lymph nodes, which provides a theoretical basis for conservative surgery. Extrafascial hysterectomy is a conservative surgical procedure that does not involve removal of parietal tissue and may be a safe and effective alternative to radical hysterectomy as an option for patients with unreserved fertility needs in early-stage, low-risk cervical cancer. In 2018, researchers used the SEER database to analyze and collect information from the period of January 1998 to December 2012 on patients who were diagnosed from January 1998 to December 2012 who were < 45 years of age with stage IB1 cervical cancer, comparing the two surgical modalities of performing non-radical excision and radical excision for cervical cancer, showed no significant difference in disease-free survival between the two groups. Thus, radical surgery did not show better oncologic outcomes compared to cervical conization, hysterectomy, or hysterectomy alone in patients with stage IB1 disease. Based on the ConCerV trial, the first multicenter prospective trial to evaluate the use of conservative surgery for early-stage, low-risk cervical cancer, the 2023 NCCN guidelines suggest that early-stage, low-risk cervical cancer should be treated with radical hand surgery if it meets the ConCerv criteria (tumor size ≤2 cm, depth of infiltration ≤10 mm, and no metastatic lesions on imaging), a conservative surgical approach is feasible, i.e, cone excision with negative margins + pelvic lymph node dissection or SLN mapping for those who will preserve fertility, and total extrafascial hysterectomy + pelvic lymph node dissection or SLN mapping for those who will not preserve fertility. In particular, at the 2023 American Society of Clinical Oncology (ASCO) Annual Meeting, an international randomized controlled phase III trial (SHAPE) initiated by the Canadian Cancer Trials Group compared the prognostic profile of patients with early-stage, low-risk cervical cancer who underwent radical hysterectomy and pelvic lymph node dissection with those who underwent hysterectomy and pelvic lymph node dissection alone, which showed that patients who underwent simple hysterectomy had a non-inferior 3-year pelvic recurrence rate to those who underwent radical hysterectomy, and that the simple hysterectomy group had a significantly lower incidence of acute adverse events and postoperative urinary retention and improved vaginal function. The above clinical trials provide strong clinical evidence for conservative surgery for early-stage, low-risk cervical cancer and have led to a series of major guideline updates as well as an expansion of our focus to conservative surgical management of patients with early-stage cervical cancer at stage 1B1 or higher.

For stage IB2 cervical cancer with tumor diameters of 2-4 cm, the current standard of care is radical hysterectomy, with a 5-year recurrence-free survival rate of 87%. An analysis of the 2018 SEER database showed that tumor lesion size ≥2 cm was an independent risk factor for disease progression, and other studies and literature reviews have shown that lesion size is one of the most important predictors of prognosis, with a statistically significantly higher risk of recurrence for lesions ≥2 cm. This may be related to the fact that larger tumor diameters simultaneously increase the proportion of vascular-positive, deep interstitial infiltration, etc., thereby increasing postoperative risk factors and the proportion of patients requiring adjuvant therapy after surgery. Thus, current guidelines only recommend non-extensive total extrafascial hysterectomy for low-risk early-stage cervical cancer, which has not been extended to patients with stage IB2, and direct conservative surgery in this population is rarely reported in the literature.

Neoadjuvant chemotherapy is commonly used in the preoperative treatment of patients with cervical cancer with local tumor diameter >4 cm. Neoadjuvant chemotherapy can reduce the size of the tumor lesion, decrease the risk of deep mesenchymal infiltration of paracervical tissue, paracervical metastasis, and positive margins for lymph node metastasis, increase the feasibility of radical surgery, and decrease the proportion of postoperative adjuvant therapy. There is increasing data to support that in patients with tumors ≥2 cm in diameter, cervical conization or radical hysterectomy after neoadjuvant chemotherapy preserves fertility and that the proportion of patients with intermediate and high risk factors requiring postoperative radiotherapy decreases significantly, with better oncologic and fertility outcomes. This also brings a new dawn for patients with stage 1B2 cervical cancer to undergo conservative surgery. With the rapid development of immunotherapy phase and treatment, the neoadjuvant treatment modality in combination with immune checkpoint inhibitors can significantly improve the EFS, pathological remission rate, etc. in numerous solid tumors. Immunotherapy has achieved remarkable results in the treatment of advanced cervical cancer, and the treatment strategy of immune checkpoint inhibitors combined with chemotherapy has become the first-line treatment for advanced or recurrent PD-L1 expression-positive cervical cancer, and Cemiplimab has been added as a preferred regimen for the second-line medication for recurrent metastatic cervical cancer in the new NCCN guideline of 2024, which is not limited to PD-L1 expression-positive population. The latest studies in cervical cancer have shown that the introduction of immunotherapy into the neoadjuvant treatment phase greatly improved the pathological remission rate of patients with locally advanced cervical cancer (IB3, IIA2 and tumor diameter ≥4cm stage IIB/IIIC1r) to 38%, and further analysis of the patients' postoperative pathological factors showed that the incision margin positivity rate was only 1. 2%, and the rate of paracervical tissue infiltration was only 2.5%, meanwhile, 69% of the neo-adjuvant immunotherapy tumor diameter ≤2 cm, and more than 50% of patients had deep mesenchymal infiltration ≤1/3. Mechanistically, more and more studies have shown that chemotherapy has an immunomodulatory effect, and chemotherapeutic agents commonly used in neoadjuvant chemotherapy for cervical cancer, including cisplatin and paclitaxel, can modulate the effector T-cell response by increasing tumor antigenicity, inducing the death of immunogenic cells, disrupting the immunosuppressive pathway, and enhancing the effector T-cell response to regulate antitumor T-cell responses. Further studies have shown that sequential administration of chemotherapy followed by immunotherapy preserves the ability of PD-L1 inhibitors to activate the immune response and may be a superior dosing strategy. Therefore, based on the application of neoadjuvant chemotherapy in conservative surgery for cervical cancer and the latest findings and theoretical basis of immunization combined with neoadjuvant chemotherapy, the investigators expect to achieve conservative surgical treatment for patients with stage IB2 cervical cancer through the application of neoadjuvant immunotherapy in stage IB2 cervical cancer by reducing the risk factors of patients to achieve therapeutic ConCerV criteria that meet the criteria for extrafascial total hysterectomy.

Cadonilimab is the world's first PD-1/CTLA-4 bispecific tumor immunotherapy that achieves immune cell activation by "double de-braking", i.e., indirectly releasing and activating immune cells by simultaneously inhibiting the two immune signaling checkpoint pathways of PD-1 and CTLA-4, thereby enhancing immune activity and strengthening the anti-tumor effect. Anti-tumor activity. Cadonilimab, the world's first new dual antibody drug for tumor immunotherapy and the first new bispecific antibody drug in China, was approved by the State Drug Administration in June 2022 for the treatment of patients with recurrent or metastatic cervical cancer who have previously failed platinum-containing chemotherapy. In the Phase II clinical trial, the anti-tumor activity of cardunculus monotherapy was encouraging and the long-term survival benefit was significant. At a median follow-up of 14.6 months, the objective remission rate of Cadonilimab monotherapy in patients with advanced cervical cancer who had failed prior platinum-containing chemotherapy was 32.3%, with 14.1% (14 cases) achieving complete remission, 18.2% (18 cases) achieving partial remission, and the median OS had not yet been reached, with an 18-month OS rate of 51.2%. In addition, Cadonilimab has demonstrated excellent efficacy and safety in clinical trials in a variety of tumors, including hepatocellular carcinoma, lung cancer and neuroendocrine tumors.

This study is an exploratory clinical trial based on recent studies of immune checkpoint inhibitors and neoadjuvant chemotherapy in patients with stage IB2 (2018 FIGO) cervical cancer, to evaluate the feasibility of extrafascial hysterectomy plus pelvic lymph node dissection in patients after Cadonilimab in combination with platinum-containing chemotherapy as neoadjuvant immunotherapy, to observe the treatment response rate, adverse effects and complications, and to assess patient survival.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosis of untreated stage IB cervical cancer with IB2 (FIGO, 2018 criteria; staging determined by two physicians of associate seniority or higher after gynecologic examination and imaging evaluation);
2. At least one measurable lesion at baseline according to RECIST 1.1 criteria, with lesion size based primarily on magnetic resonance imaging;
3. Pathologically confirmed diagnosis of cervical cancer, including cervical squamous cell carcinoma (any grade), usual type adenocarcinoma (G1 or G2 / Silva A or B), and adenosquamous carcinoma (G1 or G2);
4. Positive PD-L1 expression, Combined Positive Score (CPS) ≥1;
5. Patient age ≥18 years and ≤70 years;
6. ECOG score ≤1;
7. Laboratory tests: WBC ≥3. 5×109/L, NEU ≥1. 5×109/L, PLT ≥100×109/L, serum bilirubin ≤1.5 times the upper limit of normal, aminotransferase ≤1.5 times the upper limit of normal, and BUN and Cr ≤normal;
8. Be willing to follow up and good compliance;
9. Be willing to sign the informed consent, including compliance with the requirements and restrictions listed in the informed consent and program.

Exclusion Criteria:

1. Subjects with an active, known, or suspected autoimmune disease, or a history of an autoimmune disease, except for the following: vitiligo, alopecia areata, Graves's disease, psoriasis, or eczema that has not required systemic therapy within the last 2 years, hypothyroidism that is asymptomatic or requires only stable doses of hormone replacement therapy (due to autoimmune thyroiditis), type 1 diabetes that requires only stable doses of insulin replacement therapy, asthma that subsides completely in childhood and does not require intervention in adulthood, or diseases that do not recur in the absence of external triggers;
2. Prior treatment with immune checkpoint inhibitors, including, but not limited to, other anti-PD-1, anti-PD-L1 antibodies, CTLA-4 antibodies, or antibodies against immune co-stimulators (e.g., antibodies against ICOS, CD40, CD137, GITR, OX40 targets, etc.), or any other therapy targeting a mechanism of tumor immune action;
3. Known hypersensitivity to any component and/or any excipient of the trial prescribed medication;
4. Immunosuppressive drugs or systemic corticosteroids for immunosuppression (> 10 mg/day of prednisone or other equivalent) within 2 weeks prior to trial dosing; topical, ophthalmic, intra-articular, intranasal, and inhaled corticosteroids are permitted;
5. Received herbs with antitumor effects or drugs with immunomodulatory effects (e.g., thymidine, interferon, interleukin-2) within 2 weeks prior to the trial;
6. Active systemic infection requiring systemic treatment;
7. Serious infection within 4 weeks prior to the first dose, including but not limited to complications requiring hospitalization, sepsis, or severe pneumonia;
8. Patients with untreated chronic hepatitis B, or HBV carriers with chronic hepatitis B virus (HBV) DNA greater than 1,000 IU/mL, or patients with active hepatitis C. Inactive HBsAg carriers, patients with hepatitis B who have received treatment and are in stable condition (HBV DNA < 1000 IU/mL), and patients with cured hepatitis C are eligible for enrollment.HCV antibody-positive subjects will be eligible for the study only if they have a negative HCV RNA test;
9. Known active tuberculosis (TB), patients with suspected active TB should undergo chest X-ray and sputum examination in conjunction with clinical signs and symptoms for exclusion;
10. Immunodeficiency or human immunodeficiency virus (HIV antibody positive);
11. Subjects with active inflammatory bowel disease or a history of such disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea). Subjects who are unable to swallow or who have malabsorption syndrome, uncontrolled nausea, vomiting, diarrhea, or other gastrointestinal disorders that severely interfere with drug intake and absorption;
12. Known interstitial lung disease that is symptomatic or may interfere with detection or treatment of immune-associated pneumonia;
13. Treatment with a live or attenuated vaccine administered within 4 weeks prior to the first trial dose, inactivated seasonal influenza virus vaccine is permitted;
14. Patients who have received a prior allogeneic bone marrow transplant or solid organ transplant;
15. History of primary malignant tumor within the last 5 years;
16. Subjects who have undergone major surgery (e.g., open abdomen, open chest, organ resection, etc.) and severe trauma within 28 days prior to the first dose of the implantable infusion device is permitted;
17. Subjects with a history of gastrointestinal perforation, gastrointestinal fistula, or female genital fistula;
18. Uncontrolled other co-morbidities, symptoms, or medical history, including (i) persons with one of the following cardiovascular diseases or cardiovascular risk factors: myocardial infarction, unstable angina, pulmonary embolism, acute/continuous myocardial ischemia, cerebral vascular accident, transient ischemic attack, or other arterial or venous thrombosis, embolism, or cerebral ischemic event of clinical significance/requiring pharmacologic intervention; and persons who have had, within 6 months, a symptoms of congestive heart failure (New York Heart Association (NYHA) class III and above); (ii) clinically significant bleeding symptoms or a history of significant bleeding characteristics such as gastrointestinal bleeding, gastric ulcer bleeding, or vasculitis within 1 month prior to the first dose; (iii) clinically active hemoptysis, active diverticulitis, abdominal abscesses, and gastrointestinal obstruction; and (iv) uncontrolled pleural effusion, pericardial effusion, or ascites requiring Repeated drainage of ascites; ⑤ Abnormal liver or kidney development or history of surgery;
19. Pregnant or breastfeeding female patients; women of childbearing age who refuse to accept contraceptive measures during neoadjuvant immunotherapy;
20. Concurrent participation in other interventional clinical trials; participation in observational, non-interventional clinical trials is permitted;
21. Any condition that, in the opinion of the investigator, may result in risk in receiving the study drug or that would interfere with the evaluation of the safety of the study drug or the interpretation of the study results.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2031-01-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients meeting ConCerV criteria | 2-4 weeks after completion of neoadjuvant chemoimmunotherapy, approximately 2 years.
  Defined as the proportion (%) of all patients who met all ConCerV criteria approximately 2-4 weeks after completion of neoadjuvant chemoimmunotherapy. ConCerV criteria: no LVSI, negative margins, squamous cell carcinoma (any grade), usual type adenocarcinoma (G1 or G2 / Silva A or B) or adenosquamous carcinoma (G1 or G2), tumor size ≤2 cm, depth of infiltration ≤10 mm, no metastatic lesions seen.

SECONDARY OUTCOMES:
Objective Response Rate, ORR | 2-4 weeks after the last dose of neoadjuvant treatment and before surgery. an average of 2 years.
  the proportion of patients who had either complete response or partial response, assessed by independent central reviewers according to RECIST, version 1.1.
Proportion of patients requiring postoperative adjuvant therapy | during and after surgery; approximately 2 years
  according to the criteria for postoperative adjuvant therapy in the 2024 NCCN Guidelines, with tumor size based on size assessed by imaging prior to conization of the uterine cervix, and other pathological findings based on a combination of conization and hysterectomy results
Number of Participants with Treatment-Emergent Adverse Events as assessed by CTCAE v5.0 | Through study completion, an average of 5 year
  A treatment-emergent adverse events (TEAE) is defined as any unfavorable and unintended sign, symptom or disease temporally associated with the use of a study drug.
the surgical complication | during and after surgery; approximately 3 years
  Intraoperative bleeding, vascular injuries, bladder injuries, rectal injuries, and ureteral injuries were measured by the need for suture repair; occlusive nerve injuries were measured by complete severance, and vascular injuries required documentation of the site of injury. Postoperative complications included: cervical stenosis, cervical insufficiency, ureteral/bladder/rectal/vaginal fistula, internal hemorrhage, pelvic infection, lymphocyst, lymphatic fistula, lower extremity edema, lower extremity venous thrombosis, urinary retention, nerve injury, and bowel obstruction.
Pathologic Complete Response | during the surgery; approximately 2 years.
  Pathologic complete response (PCR) refers to the absence of invasive/in situ cancer and/or lymph nodes
Overall survival, OS | the time from randomization to death. A total of 7 years.
  as the time from randomization to death
progression-free survival, PFS | Until 5 years after the last case enrollment. a total of 7 years.
  the chances of staying free of disease progression for patients with cervical cancer.
Time to successful postoperative urinary catheter removal, rate of urinary retention and incontinence | Until the end of this study, A total of 7 years.
  Time to successful postoperative urinary catheter removal: The time from the date of surgery to the date when the urinary catheter is removed and no longer needs to be reinserted.
  Urinary retention: Urinary retention was defined as the patient's inability to urinate successfully, defined as a residual urine volume of ≥100 mL in the bladder as determined by ultrasound after urinary catheter removal, or inability to urinate independently requiring reintroduction of a urinary catheter.
  Urinary incontinence: The presence of urinary incontinence was determined by history and physical examination.
Patient Reported Outcomes | assessed at baseline, before cone biopsy, 1 week after hysterectomy (1 week after the end of adjuvant therapy if participants have), every time participants follow-up. A total of 7 years.
  1. Quality of Life questionnaire (composed of the QLQ-C30, QLQ-CX24); 2. Sexual Health questionnaire (composed of the FSFI); 3. Health Economics questionnaire (composed of the EQ-5D)

CONTACTS AND LOCATIONS:
Overall Officials: Ding Ma, Study Chair — Tongji Hospital
Locations (2):
- China (2):
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Qilu Hospital of Shandong University, Jinan, Shandong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hu Y, Cheng H, Chen J, Chen S, Han Y, Sun C, Chen G, Li K. Neoadjuvant chemotherapy plus cadonilimab followed by extra-fascial hysterectomy for International Federation of Gynecology and Obstetrics stage IB2 cervical cancer: a prospective, multi-center, single-arm, phase 2 trial. Int J Gynecol Cancer. 2026 Jan 5:104457. doi: 10.1016/j.ijgc.2025.104457. Online ahead of print. PMID 41582028